CLINICAL TRIAL: NCT01006096
Title: Phase II Randomized, Double-blind, Placebo-controlled, Two-arm Study to Evaluate the Safety and Efficacy of Erlotinib in the Treatment of Moderate to Severe Psoriasis
Brief Title: Erlotinib for Treatment of Psoriasis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: IND not obtained
Sponsor: Northwestern University (Other)
Collaborators: OSI Pharmaceuticals (Industry)
Responsible Party: Anne E. Laumann, MBChB, MRCP (UK)/Associate Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MEL-041509
Record Dates: First submitted 2009-10-29; First posted 2009-11-02 (Estimated); Last update posted 2014-11-10 (Estimated); Status verified 2014-11

CONDITIONS: Psoriasis
Keywords: Psoriasis; double-blind; randomized; placebo-controlled; erlotinib; efficacy
MeSH Terms: conditions — Psoriasis | interventions — Erlotinib Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Erlotinib (Experimental)
  Interventions: Drug: erlotinib
- Placebo tablets (Placebo Comparator)
  Interventions: Other: placebo tablet

INTERVENTIONS:
Drug: erlotinib — 100mg tablet, once daily for 16 weeks
  Other Names: Tarceva
  Arms: Erlotinib
Other: placebo tablet — placebo tablet (lactose), once daily for 16 weeks
  Arms: Placebo tablets

SUMMARY:
The purpose of this study is to determine whether erlotinib is effective in the treatment of psoriasis.

DETAILED DESCRIPTION:
Psoriasis vulgaris is a disease that affects 25 million people in North America and Europe. It often presents in late adolescence and usually persists for life. Current therapies target specific immune molecules that are implicated in the cause of this disease. For example, biologic agents that are used in severe psoriasis are aimed at inflammatory mediators. These therapies have been proven to be effective but also have their limitations.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of moderate to severe psoriasis
* Must have documented moderate to severe psoriasis by the Physician's Global Assessment (PGA) and the Psoriasis Area Severity Index (PASI)
* Must be able to swallow tablets
* Must be able to provide written informed consent
* Subjects with reproductive potential (menopausal for less than 1 year and not surgically sterilized) must practice effective contraceptive measures throughout the study and thirty days after discontinuation of study drug. Women of childbearing potential must provide negative pregnancy test (serum or urine) within 14 days prior to randomization.

Exclusion Criteria:

* Use of concurrent agents/therapies for psoriasis
* Bilirubin > 3 X ≥ ULN or moderate to severe hepatic impairment
* Pregnant or breast-feeding females
* Subjects currently receiving other anticancer treatments
* Subjects currently receiving other biologic treatments
* Subjects currently receiving blood thinners (warfarin or heparin)
* Subjects who currently smoke
* Subjects with other skin disease which in the opinion of the investigator, would inhibit the ability to use the PGA and PASI evaluation methods

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
To determine efficacy of erlotinib in treatment of moderate to severe psoriasis measured by the Psoriasis Area and Severity Index (PASI) and the Physician's Global Assessment (PGA). | week 4, 8, 12, 16, and 24

SECONDARY OUTCOMES:
To determine the rate of dose reduction or interruption as a result of adverse events. | week 4, 8, 12, 16, and 24
To determine quality of life using the Dermatology Life Quality Index (DLQI). | week 4, 8, 12, 16, and 24

CONTACTS AND LOCATIONS:
Overall Officials: Anne E Laumann, MBChB, MRCP (UK), Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Feinberg School of Medicine Department of Dermatology, Chicago, Illinois, United States

REFERENCES:
- [Background] Lowes MA, Bowcock AM, Krueger JG. Pathogenesis and therapy of psoriasis. Nature. 2007 Feb 22;445(7130):866-73. doi: 10.1038/nature05663. PMID 17314973
- [Background] Shepherd FA, Rodrigues Pereira J, Ciuleanu T, Tan EH, Hirsh V, Thongprasert S, Campos D, Maoleekoonpiroj S, Smylie M, Martins R, van Kooten M, Dediu M, Findlay B, Tu D, Johnston D, Bezjak A, Clark G, Santabarbara P, Seymour L; National Cancer Institute of Canada Clinical Trials Group. Erlotinib in previously treated non-small-cell lung cancer. N Engl J Med. 2005 Jul 14;353(2):123-32. doi: 10.1056/NEJMoa050753. PMID 16014882
- [Background] Lacouture ME. Mechanisms of cutaneous toxicities to EGFR inhibitors. Nat Rev Cancer. 2006 Oct;6(10):803-12. doi: 10.1038/nrc1970. PMID 16990857
- [Background] Wierzbicka E, Tourani JM, Guillet G. Improvement of psoriasis and cutaneous side-effects during tyrosine kinase inhibitor therapy for renal metastatic adenocarcinoma. A role for epidermal growth factor receptor (EGFR) inhibitors in psoriasis? Br J Dermatol. 2006 Jul;155(1):213-4. doi: 10.1111/j.1365-2133.2006.07299.x. No abstract available. PMID 16792781
- [Background] Ben-Bassat H, Vardi DV, Gazit A, Klaus SN, Chaouat M, Hartzstark Z, Levitzki A. Tyrphostins suppress the growth of psoriatic keratinocytes. Exp Dermatol. 1995 Apr;4(2):82-8. doi: 10.1111/j.1600-0625.1995.tb00227.x. PMID 7640880
- [Background] Powell TJ, Ben-Bassat H, Klein BY, Chen H, Shenoy N, McCollough J, Narog B, Gazit A, Harzstark Z, Chaouat M, Levitzki R, Tang C, McMahon J, Shawver L, Levitzki A. Growth inhibition of psoriatic keratinocytes by quinazoline tyrosine kinase inhibitors. Br J Dermatol. 1999 Nov;141(5):802-10. doi: 10.1046/j.1365-2133.1999.03152.x. PMID 10583160
- [Background] Ben-Bassat H, Klein BY. Inhibitors of tyrosine kinases in the treatment of psoriasis. Curr Pharm Des. 2000 Jun;6(9):933-42. doi: 10.2174/1381612003400182. PMID 10828317
- [Background] Ben-Bassat H, Levitzki A. Inhibitors of tyrosine kinases in the treatment of psoriasis. Isr Med Assoc J. 2000 Jul;2 Suppl:69-73. No abstract available. PMID 10909421
- [Background] Halin C, Fahrngruber H, Meingassner JG, Bold G, Littlewood-Evans A, Stuetz A, Detmar M. Inhibition of chronic and acute skin inflammation by treatment with a vascular endothelial growth factor receptor tyrosine kinase inhibitor. Am J Pathol. 2008 Jul;173(1):265-77. doi: 10.2353/ajpath.2008.071074. Epub 2008 Jun 5. PMID 18535184
- [Background] Forsberg S, Ostman A, Rollman O. Regeneration of human epidermis on acellular dermis is impeded by small-molecule inhibitors of EGF receptor tyrosine kinase. Arch Dermatol Res. 2008 Oct;300(9):505-16. doi: 10.1007/s00403-008-0853-2. Epub 2008 Apr 30. PMID 18446355
- [Background] Neyns B, Meert V, Vandenbroucke F. Cetuximab treatment in a patient with metastatic colorectal cancer and psoriasis. Curr Oncol. 2008 Aug;15(4):196-7. doi: 10.3747/co.v15i4.228. PMID 18769609
- [Background] Trivin F, Boucher E, Raoul JL. Complete sustained regression of extensive psoriasis with cetuximab combination chemotherapy. Acta Oncol. 2004;43(6):592-3. doi: 10.1080/02841860410020211. No abstract available. PMID 15370619